CLINICAL TRIAL: NCT01458938
Title: Substance P Neuropeptide Levels in Saliva, Serum and Cerebrospinal Fluid in Patients With Spinal Disease: A Pilot Study
Brief Title: This Study is to Determine if Degenerative Spinal Pain and Disorders Cause the Levels of Substance P to Change in a Patients Saliva, Blood and/or Cerebrospinal Fluid.
Acronym: Substance P
Status: Terminated | Type: Observational
Why Stopped: Study will need to be redesigned for improved efficacy.
Sponsor: Carolina Neurosurgery & Spine Associates (Other)
Responsible Party: Sponsor
Other Study IDs: Substance P
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Disease; Spinal Radiculopathy; Myelopathy; Neurogenic Claudication
MeSH Terms: conditions — Spinal Diseases; Spinal Cord Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, saliva and cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Healthy volunteers
- surgery for spinal radiculopathy
  Interventions: Other: treatment plan
- surgery for axial spine pain
  Interventions: Other: treatment plan
- myelography for spinal pain
  Interventions: Other: treatment plan

INTERVENTIONS:
Other: treatment plan — Data Collection Study
  Groups: myelography for spinal pain; surgery for axial spine pain; surgery for spinal radiculopathy

SUMMARY:
The objective of this pilot study is to determine if degenerative spinal disorders such as acute radiculopathy, myelopathy, stenosis, or disc and facet disease cause detectable alterations in Substance P levels in saliva, serum and cerebrospinal fluid. If this pilot study shows a correlation between Substance P levels and pain associated with degenerative spinal disorders, then a larger study will be initiated to determine the feasibility of using Substance P levels in the diagnosis and treatment of degenerative spinal disease.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing spinal surgery for medically refractory spinal radiculopathy,
* myelopathy or neurogenic claudication based on either history, physical examination or radiologic studies demonstrating neural compression or degenerative disc disease.
* Undergoing surgery for medically refractory axial spinal pain.

Exclusion Criteria:

* Previous spinal procedures or operations,
* radicular pain,
* history of fibromyalgia,
* chronic pain,
* rheumatoid arthritis,
* autoimmune disorders,
* HIV,
* PTSD,
* Major Depressive Disorder,
* migraine headaches or active rhinosinusitis,
* nicotine intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2009-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Substance P Neuropeptide Levels in Saliva And Serum in Patients with Spinal Disease: A Pilot Study | 2009-2014
  Study was closed pending re-design at some future date to improve efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Deshmukh, M.D., Principal Investigator — Carolina Neurosurgery & Spine Associates
Locations (1):
- Carolina Neurosurgery and Spine Associates, P.A., Charlotte, North Carolina, United States